CLINICAL TRIAL: NCT01930370
Title: Effect of Varied Dialysate Bicarbonate Levels on Phosphate and Potassium Removal: A Pilot Study
Brief Title: Effect of Varied Dialysate Bicarbonate Levels on Phosphate and Potassium Removal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Elizabeth Harvey, Project Investigator, The Hospital for Sick Children
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1000014657
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Dialysis Patients
Keywords: pediatrics; phosphate and postassium revmoval; dialysate bicarbonate modeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hemodialysis patients (Experimental): Each patient will be evaluated during a total of 3.5 weeks correlating to routine dialysis treatment appointments. Each participant will start with low bicarbonate, followed by the washout phase (standard bicarbonate), then high bicarbonate, finishing with the follow up period. Dialysis prescription is standardized for each patient throughout the entire 3.5 week study period.
  Interventions: Drug: Bicarbonate hemodialysis solution (low concentration); Drug: Bicarbonate hemodialysis solution (high concentration)

INTERVENTIONS:
Drug: Bicarbonate hemodialysis solution (low concentration) — One-week experimental session (3 dialysis treatments) with low dialysate bicarbonate (28 mmol/L)
Drug: Bicarbonate hemodialysis solution (high concentration) — One-week experimental session with high dialysate bicarbonate (38 mmol/L)

SUMMARY:
Modeling of bicarbonate within the dialysate fluid, specifically a lower than standard concentration has been suggested in facilitating the removal of phosphate and potassium. To test this hypothesis, the study will use a cross-over study design to evaluate phosphate and potassium removal during dialysis by altering bicarbonate concentration in dialysis fluid (i.e. high bicarbonate, standard bicarbonate washout, low bicarbonate), and compare the effects of the different dialysate bicarbonate concentrations on the removal of phosphate and potassium during hemodialysis

DETAILED DESCRIPTION:
Elevation of blood phosphate levels in chronic dialysis patients is associated with increased mortality due to cardiovascular events, and if sustained leads to hyperactivity of parathyroid glands and renal bone disease. Similarly, increased calcium-phosphate product as a result of elevated levels of phosphate in the blood is an additional risk factor for vascular calcification. Elevated blood potassium levels is another major electrolyte disorder in patients with advanced renal disease which is potentially life threatening. Therefore control of blood phosphate and potassium levels is a fundamental component of treatment for end stage renal disease. Management of hyperelectrolyte levels in renal failure patients requires restriction of phosphate and potassium intake through dietary measures, promotion of excretion via GI tract through medication delivery (i.e. supplementary binders), and removal through dialysis. All these strategies come with limitations however, specifically adherence to dietary restrictions and medication compliance is poor due to lack of immediate repercussions, as well as the complex kinetics involved with removal via dialysis given the dependence on duration and frequency of dialysis whose manipulation is limited by time considerations for the patient and scheduling issues in the dialysis unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients 0-18 years old
* Patients receiving maintenance hemodialysis* for a total of 9-15 hours per week
* Pre-dialysis serum potassium value between 4.0 and 6.5 mmol/L on the first day of the treatment protocol
* Pre-dialysis serum phosphate value greater than low normal for age on the first day of the treatment protocol
* Pre-dialysis serum bicarbonate (total CO2) value between 18 and 30 mmol/L on the first day of the treatment protocol
* Pre-dialysis corrected calcium value between 1.80-2.85 mmol/L on the first day of the treatment protocol

Exclusion Criteria:

* Hemodynamically unstable patients (requiring inotropes or midodrine for support).
* Pre-dialysis potassium value < 4.0 or > 6.5 mmol/L on the first day of the treatment protocol
* Pre-dialysis serum phosphate value less than low normal for age on the first day of the treatment protocol (i.e. hypophosphatemia)
* Pre-dialysis serum bicarbonate (total CO2) value <18 or > 30 mmol/L on the first day of the treatment protocol
* Pre-dialysis corrected calcium <1.8 and >2.85 mmol/L on the first day of the treatment protocol
* Patients mechanically ventilated
* Drugs that could modify internal phosphate and potassium balance such as insulin, bicarbonate injection, hypertonic dextrose solution or mannitol infusion during HD

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Phosphate/Potassium Removal | Dialysis Treatment 1 (Day 1) - Pre and Post dialysis (0hrs and 4hours)
  The amount of phosphate/potassium removed with each dialysis as measured from dialysate aliquots and total calculated volume of dialysate. The following formula will be used to calculate Phosphate (PO4) and Potassium (K) mass removal (mmol/treatment):
  Calculation based on the concentration of K/PO4 (mmol/L) in dialysate x (calculated volume of dialysate + calculated volume of ultrafiltrate)
Phosphate/Potassium Removal | Dialysis Treatment 2 (Day 2) - Pre and Post dialysis (0hrs and 4hours)
  The amount of phosphate/potassium removed with each dialysis as measured from dialysate aliquots and total calculated volume of dialysate. The following formula will be used to calculate Phosphate (PO4) and Potassium (K) mass removal (mmol/treatment):
  Calculation based on the concentration of K/PO4 (mmol/L) in dialysate x (calculated volume of dialysate + calculated volume of ultrafiltrate)
Phosphate/Potassium Removal | Dialysis Treatment 3 (Day 3) - Pre and Post dialysis (0hrs, 4hours, 5hours)
  The amount of phosphate/potassium removed with each dialysis as measured from dialysate aliquots and total calculated volume of dialysate. The following formula will be used to calculate Phosphate (PO4) and Potassium (K) mass removal (mmol/treatment):
  Calculation based on the concentration of K/PO4 (mmol/L) in dialysate x (calculated volume of dialysate + calculated volume of ultrafiltrate)
Phosphate/Potassium Removal | Dialysis Treatment 7 (Day 15) - Pre and Post dialysis (0hrs, 4hours)
  The amount of phosphate/potassium removed with each dialysis as measured from dialysate aliquots and total calculated volume of dialysate. The following formula will be used to calculate Phosphate (PO4) and Potassium (K) mass removal (mmol/treatment):
  Calculation based on the concentration of K/PO4 (mmol/L) in dialysate x (calculated volume of dialysate + calculated volume of ultrafiltrate)
Phosphate/Potassium Removal | Dialysis Treatment 8 (Day 16) - Pre and Post dialysis (0hrs, 4hours)
  The amount of phosphate/potassium removed with each dialysis as measured from dialysate aliquots and total calculated volume of dialysate. The following formula will be used to calculate Phosphate (PO4) and Potassium (K) mass removal (mmol/treatment):
  Calculation based on the concentration of K/PO4 (mmol/L) in dialysate x (calculated volume of dialysate + calculated volume of ultrafiltrate)
Phosphate/Potassium Removal | Dialysis Treatment 9 (Day 17) - Pre and Post dialysis (0hrs, 4hours, 5hours)
  The amount of phosphate/potassium removed with each dialysis as measured from dialysate aliquots and total calculated volume of dialysate. The following formula will be used to calculate Phosphate (PO4) and Potassium (K) mass removal (mmol/treatment):
  Calculation based on the concentration of K/PO4 (mmol/L) in dialysate x (calculated volume of dialysate + calculated volume of ultrafiltrate)

SECONDARY OUTCOMES:
Plasma Phosphate Levels | Baseline and Post Dialysis (4hours)
  Measurement of the biochemical (serum) parameters of Phosphate for each dialysis treatment
Plasma Potassium Levels | Pre and Post Dialysis
  Measurement of the biochemical (serum) parameters of Potassium for each dialysis treatment
Total Plasma CO2 (bicarbonate) | Pre and Post Dialysis (0 and 4hours)
  Measurement of the biochemical (serum) parameters of CO2 (bicarbonate) for each dialysis treatment
Corrected Calcium Measurement | Pre and Post Dialysis (0 and 4hours)
  Biochemical measurement of the blood for corrected caclium (calcium and albumin) for each dialysis treatment
Dialysis Adequacy (Kt/ V) | Pre and Post Dialysis (0 and 4hours)
  Measurement of Blood urea will be performed for each dialysis treatment.
Dialysis Adequacy (Urea Reduction Ratio -URR) | Pre and Post Dialysis (0 and 4hours)
  Measurement of Blood urea will be performed for each dialysis treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Geary, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada